CLINICAL TRIAL: NCT00041470
Title: Navelbine, Taxol, Herceptin and Neupogen in Stage IV Breast Cancer: A Phase I - II Trial
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor withdrew the study
Sponsor: University of Washington (Other)
Collaborators: Amgen (Industry); Bristol-Myers Squibb (Industry); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Julie Ruth Gralow, Professor of Medicine, Medicine/Oncology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18245
Record Dates: First submitted 2002-07-09; First posted 2002-07-10 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Vinorelbine; Trastuzumab; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Weekly paclitaxel, vinorelbine and GCSF (Experimental): Weekly paclitaxel (50 mg/m2 IV) and weekly vinorelbine (20 mg/m2 IV) with daily G-CSF support and Herceptin for patients with HER-2/neu positive disease.
  Paclitaxel weekly. Dose levels:
  50 mg/m2, 60 mg/m2, 70 mg/m2, 80 mg/m2
  Vinorelbine (Navelbine) administered one hour after paclitaxel, weekly. Dose levels:
  20 mg/m2, 22.5 mg/m2, 25 mg/m2, 27.5 mg/m2
  Patients who are HER-2+ and IV infusion. Herceptin 4 mg/kg IV given only on day 1 of the first cycle. Herceptin 2 mg/kg IV, maintenance dose will be given every week starting with week 2.
  G-CSF (filgrastim, Neupogen) 5 mg/kg/day s.c., administered daily
  Interventions: Drug: Paclitaxel; Drug: Vinorelbine; Drug: Herceptin; Drug: Filgrastim

INTERVENTIONS:
Drug: Paclitaxel — 50 mg/m2 IV weekly. Treatment continues until disease progression, excessive toxicity or other reason to remove the patient from protocol treatment.
  Other Names: Taxol
Drug: Vinorelbine — 20 mg/m2 IV weekly. Treatment continues until disease progression, excessive toxicity or other reason to remove the patient from protocol treatment.
  Other Names: Navelbine
Drug: Herceptin — 4 mg/kg IV loading dose day 1 of first week followed by 2 mg/kg IV maintenance dose on each subsequent week. Treatment continues until disease progression, excessive toxicity or other reason to remove the patient from protocol treatment.
  Other Names: Trastuzumab
Drug: Filgrastim — 5 mcg/kg daily including the day of IV chemotherapy. Treatment continues until disease progression, excessive toxicity or other reason to remove the patient from protocol treatment.
  Other Names: G-CSF; Neupogen

SUMMARY:
The purposes of this are:

* To determine the highest doses of Taxol and Navelbine that we can safely give to patients;
* To determine what kind of side effects are caused by the combination of Taxol, Navelbine and G-CSF;
* To determine whether the combination of Taxol, Navelbine and G-CSF is more effective than standard therapy in treating metastatic breast cancer and prolonging life;

DETAILED DESCRIPTION:
Complete response (CR) in advanced breast cancer is an important predictor of improved survival. The largest experience reported with long-term follow-up in this regard is from M.D. Anderson Hospital, with a median survival of 33 months and 5-year survival of 19% among patients who achieved a CR with doxorubicin-based chemotherapy.19 We believe that our institutional experience to date indicates that CR rates in excess of 20% can be achieved in second-line chemotherapy from the combination of vinorelbine and a taxane, provided that G-CSF is given. For the reasons outlined, we believe that dose density is likely to be important for both classes of agents, but dose intensity may be most important for vinorelbine. Both paclitaxel and docetaxel can be given on a weekly schedule with some success, but it appears that myelosuppression is a more frequent dose-limiting toxicity on this schedule for docetaxel. For the current trial, we therefore propose to study weekly paclitaxel in combination with dose-intensive vinorelbine, utilizing continuous G-CSF support as in our prior studies. We believe that starting doses of 60 mg/m2 for paclitaxel and 20 mg/m2 for vinorelbine will be well tolerated, but our experience to date, treating 3 patients off study at these doses without G-CSF support, indicates that some will require G-CSF even at this dose level: we observed grade 4 neutropenia in 2 of the 3. Our intention in this trial is to determine the optimal dose of these two agents when continuous growth factor support is provided. We will be starting at a ratio of 0.8 for vinorelbine and 0.75 for paclitaxel (assuming 80 mg/m2/week as a "full" dose for the later agent).

It is now widely appreciated that patients with metastatic breast cancer whose tumors over express HER-2-neu demonstrate benefit from the addition of trastuzumab (Herceptin) to a chemotherapy program with paclitaxel as a single agent.20 Such patients will be allowed to receive trastuzumab in the standard dose and schedule (4 mg/kg loading dose, then 2 mg/kg/week) given IV, in addition to paclitaxel and vinorelbine. Since trastuzumab does not produce myelosuppression or neuropathy (the anticipated dose-limiting toxicities for vinorelbine and paclitaxel, respectively), and neither of these agents combined separately with trastuzumab produces unusual or severe new side effects, this should not affect the dose escalation scheme for the chemotherapeutic agents.

ELIGIBILITY:
PATIENT ELIGIBILITY

Inclusion Criteria:

* Patient has stage IV, microscopically-confirmed carcinoma of the breast with histologic slides and/or blocks available for review.
* Patient has had one or less prior regimens for metastatic disease. Prior paclitaxel by 3, 24 or 96-hour infusion is permitted as long as it did not result in any neuropathy. Prior docetaxel on an every 3-week schedule is permitted.
* Measurable (bidimensionally) or evaluable disease.
* Age > 18.
* Karnofsky Performance Status > 70% (ECOG, < 2) at screen and on the first day of treatment.
* Life expectancy > 16 weeks.
* Prior irradiation is permitted, provided:
* Prior irradiation does not exceed 25% of the estimated bone marrow volume. (See Appendix I)
* Measurable/evaluable disease must exist outside the radiation field OR there must be histologic proof of progressive disease within a radiation field.
* Informed consent must be obtained prior to registration.
* Patients must be > 2 weeks from prior surgery; > 3 weeks from radiation therapy to the pelvis, spine or long bones; > 3 weeks from prior chemotherapy (> 6 weeks for mitomycin C or nitrosureas), or > 2 weeks from prior hormonal therapy.
* All patients must have placement of appropriate central venous access device.
* Tumor HER2/neu expression must be determined prior to study enrollment. Assessment may be by fluorescence in situ hydridization (FISH) assay or by immunohistochemistry (ICC). If determination is intermediate by ICC, FISH must be performed. For enrollment purposes, the phase I portion of the study will not discriminate based on HER2 status. However, documentation of patients' HER2 status will be maintained and Herceptin will be prescribed for all HER2 positive patients. The phase II portion of the study will enroll 30 patients who are documented HER2 overexpressors and 30 patients who are non-overexpressors.

Exclusion Criteria:

* Granulocytes < 1,500/mm3.
* Platelets < 100,000/mm3.
* Hemoglobin < 9 gm/dl.
* Creatinine > 2.0 mg/dl.
* Total bilirubin > 2 mg/dl.
* Visceral crisis characterized by rapidly progressive hepatic or lymphangitic lung metastases.
* Medically unstable as judged by the patient's physician.
* Pregnancy or lactation; failure to employ adequate contraception.
* Uncontrolled CNS disease.
* Pre-existing clinically significant peripheral neuropathy except for abnormalities due to cancer.
* Psychological, familial, sociological or geographical conditions which do not permit weekly medical follow-up and compliance with the study protocol.
* Prior therapy with vinorelbine or prior therapy with a taxane that resulted in neuropathy.
* Known hypersensitivity to E. coli-derived proteins, Filgrastim, or any component of the product as Neupogen® is contraindicated in such subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2001-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie R. Gralow, M.D., Principal Investigator — University of Washington
Locations (1):
- Seattle Cancer Care Alliance, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Paclitaxel, Vinorelbine, G-CSF, Herceptin - no Placebo: Weekly paclitaxel (50 mg/m2 IV) and weekly vinorelbine (20 mg/m2 IV) with daily G-CSF support and Herceptin for patients with HER-2/neu positive disease. Treatment continues until disease progression, toxicity or other reason to remove the patient from protocol treatment.
  Paclitaxel is administered weekly. Dose levels:
  50 mg/m2, 60 mg/m2, 70 mg/m2, 80 mg/m2
  Vinorelbine (Navelbine) is administered one hour after paclitaxel, every week. Dose levels:
  20 mg/m2, 22.5 mg/m2, 25 mg/m2, 27.5 mg/m2
  Patients whose tumors over express HER-2-neu and who meet the cardiac safety criteria will receive weekly Herceptin administered by intravenous infusion.
  Herceptin 4 mg/kg IV given only on day 1 of the first cycle. Herceptin 2 mg/kg IV, maintenance dose will be given every week starting with week 2.
  G-CSF (filgrastim, Neupogen) 5 mg/kg/day s.c., is administered daily including the day of chemotherapy.
  Paclitaxel: 50 mg/m2 IV weekly. Treatment continues until progression
Period: Overall Study
Arm/Group | Paclitaxel, Vinorelbine, G-CSF, Herceptin - no Placebo
Started | 38
Completed | 0
Not Completed | 38
Not completed — Loss of Funding | 38

BASELINE CHARACTERISTICS:
Groups:
- Phase I/II: Weekly paclitaxel (50 mg/m2 IV) and weekly vinorelbine (20 mg/m2 IV) with daily G-CSF support and Herceptin for patients with HER-2/neu positive disease. Treatment continues until disease progression, toxicity or other reason to remove the patient from protocol treatment.
  Paclitaxel is administered weekly. Dose levels:
  50 mg/m2, 60 mg/m2, 70 mg/m2, 80 mg/m2
  Vinorelbine (Navelbine) is administered one hour after paclitaxel, every week. Dose levels:
  20 mg/m2, 22.5 mg/m2, 25 mg/m2, 27.5 mg/m2
  Patients whose tumors over express HER-2-neu and who meet the cardiac safety criteria will receive weekly Herceptin administered by intravenous infusion.
  Herceptin 4 mg/kg IV given only on day 1 of the first cycle. Herceptin 2 mg/kg IV, maintenance dose will be given every week starting with week 2.
  G-CSF (filgrastim, Neupogen) 5 mg/kg/day s.c., is administered daily including the day of chemotherapy.
  Paclitaxel: 50 mg/m2 IV weekly. Treatment continues until disease pr
Arm/Group | Phase I/II
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 46.5 [27 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 0
Baseline Participants [Number; unit: participants] | 38

OUTCOME MEASURES:

1. Primary Outcome: To Measure Response Rates, Time to Progression and Survival in Patients so Treated.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Weekly Paclitaxel, Vinorelbine and GCSF: Weekly paclitaxel (50 mg/m2 IV) and weekly vinorelbine (20 mg/m2 IV) with daily G-CSF support and Herceptin for patients with HER-2/neu positive disease.
  Paclitaxel weekly. Dose levels:
  50 mg/m2, 60 mg/m2, 70 mg/m2, 80 mg/m2
  Vinorelbine (Navelbine) administered one hour after paclitaxel, weekly. Dose levels:
  20 mg/m2, 22.5 mg/m2, 25 mg/m2, 27.5 mg/m2
  Patients who are HER-2+ and IV infusion. Herceptin 4 mg/kg IV given only on day 1 of the first cycle. Herceptin 2 mg/kg IV, maintenance dose will be given every week starting with week 2.
  G-CSF (filgrastim, Neupogen) 5 mg/kg/day s.c., administered daily
  Paclitaxel: 50 mg/m2 IV weekly. Treatment continues until disease progression, excessive toxicity or other reason to remove the patient from protocol treatment.
  Vinorelbine: 20 mg/m2 IV weekly. Treatment continues until disease progression, excessive toxicity or other reason to remove the patient from protocol treatment.
  Herceptin: 4 mg/kg IV loading dose day 1
Arm/Group | Weekly Paclitaxel, Vinorelbine and GCSF
Number analyzed (Participants) | 38
Participants
  Complete Response | 6
  Partial Response | 14
  Stable Disease | 9
  Progressive Disease | 8
  Inevaluable | 1

2. Secondary Outcome: To Measure the Qualitative and Quantitative Toxicity of This Regimen.
Time Frame: <=18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Weekly Paclitaxel, Vinorelbine and GCSF
Number analyzed (Participants) | 38
Participants
  >=Grade 3 Toxicity | 30
  serious adverse events | 10

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Weekly Paclitaxel and Vinorelbine With GCSF Support: Weekly paclitaxel (50 mg/m2 IV) and vinorelbine (20 mg/m2 IV) with daily G-CSF and Herceptin for patients with HER-2+ disease. Treatment until disease progression, excessive toxicity or other reason to remove the patient from protocol treatment.
  Paclitaxel administered weekly. Dose levels:
  50 mg/m2, 60 mg/m2, 70 mg/m2, 80 mg/m2
  Vinorelbine (Navelbine) administered one hour after paclitaxel, weekly. Dose levels:
  20 mg/m2, 22.5 mg/m2, 25 mg/m2, 27.5 mg/m2
  Patients who are HER-2+ and meet the cardiac safety criteria will receive weekly Herceptin administered by infusion.
  Herceptin 4 mg/kg IV given only on day 1 of the first cycle. Herceptin 2 mg/kg IV, maintenance dose will be given every week starting with week 2.
  G-CSF (filgrastim, Neupogen) 5 mg/kg/day s.c., is administered daily including the day of chemotherapy.
  Paclitaxel: 50 mg/m2 IV weekly. Treatment continues until disease pr
Arm/Group | Weekly Paclitaxel and Vinorelbine With GCSF Support
Serious Adverse Events (participants affected / at risk) | 10/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weekly Paclitaxel and Vinorelbine With GCSF Support (N=38)
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 4 (4)
Mucositis (Infections and infestations) | 2 (2) — Requiring total parenteral nutrition
Congestive Heart Failure (Cardiac disorders) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weekly Paclitaxel and Vinorelbine With GCSF Support (N=38)
Neutropenia (Blood and lymphatic system disorders) | 20 (20)
Thrombocytopenia (Blood and lymphatic system disorders) | 16 (16)
Vomiting (Gastrointestinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No